CLINICAL TRIAL: NCT01605877
Title: Clinical Investigation of AcrySof® IQ ReSTOR® Multifocal Intraocular Lens Model SN6AD2
Brief Title: AcrySof® IQ ReSTOR® +2.5 D Multifocal Intraocular Lens (IOL) Model SN6AD2 [SV25T0] in Japan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J-11-037
Record Dates: First submitted 2012-05-22; First posted 2012-05-25 (Estimated); Results first posted 2015-06-09 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-06

CONDITIONS: Cataracts
Keywords: Cataracts; Intraocular lens; Multifocal; Presbyopia
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SN6AD2 (Experimental): AcrySof® IQ ReSTOR® +2.5 D Multifocal IOL Model SN6AD2 [SV25T0], bilateral implantation
  Interventions: Device: AcrySof® IQ ReSTOR® +2.5 D Multifocal IOL Model SN6AD2 [SV25T0]

INTERVENTIONS:
Device: AcrySof® IQ ReSTOR® +2.5 D Multifocal IOL Model SN6AD2 [SV25T0] — Multifocal IOL with extended secondary focal point implanted for long-term use over the lifetime of the cataract patient

SUMMARY:
The purpose of this study is to evaluate safety and effectiveness of AcrySof® IQ ReSTOR® +2.5 D Multifocal IOL Model SN6AD2 [SV25T0] in Japanese cataract patients.

DETAILED DESCRIPTION:
Each subject completed a preoperative examination of both eyes, implantation of IOL at the operative visit for each eye, and up to 8 postoperative visits (each eye examined at Day 1-2, Day 7-14, and Day 30-60, with binocular visits at Day 120-180 and Day 330-420 after the second implantation). The second implantation occurred within 30 days of the first.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent;
* Diagnosed with bilateral cataracts;
* Planned cataract removal by phacoemulsification;
* Potential postoperative visual acuity of 0.5 decimal or better in both eyes;
* Preoperative astigmatism ≤ 1.5 diopter;
* Clear intraocular media other than cataract in study eyes;
* Calculated lens power within the available range;
* Able to undergo second eye surgery within 30 days of the first eye surgery;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Significant irregular corneal aberration as demonstrated by corneal topography;
* Any inflammation or edema (swelling) of the cornea;
* Diagnosed degenerative visual disorders predicted to cause future acuity losses to a level worse than 0.5 decimal;
* Diabetic retinopathy;
* Previous refractive surgery, retinal detachment, corneal transplant;
* Glaucoma;
* Pregnancy;
* Currently participating in another investigational drug or device study;
* Exclusion criteria during surgery;
* Other protocol-defined exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Kodama, Study Director — Alcon Japan, Ltd.
Locations (2):
- Japan (2):
  - Hayashi Eye Hospital, Fukuoka, Fukuoka
  - Tokyo Dental College Suidobashi Hospital, Chiyoda-ku, Tokyo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 2 study sites located in Japan.
Pre-assignment Details: Of the 70 subjects enrolled, 6 were discontinued prior to first implantation due to withdrawn consent (1) and meeting exclusion criteria (5). This reporting group includes all implanted subjects (64).
Period: Overall Study
Arm/Group | SN6AD2
Started | 64
Completed | 63
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all implanted subjects.
Arm/Group | SN6AD2
Number analyzed (Participants) | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (7.2)
Age, Customized [Number; unit: participants]
  <60 years | 10
  60-69 years | 29
  70-79 years | 24
  ≥ 80 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 23
Region of Enrollment [Number; unit: participants]
  Japan | 64

OUTCOME MEASURES:

1. Primary Outcome: Uncorrected Decimal VA (5 m)
Description: Visual acuity (VA) was tested monocularly (each eye separately) at all visits and binocularly (both eyes together) at Day 30-60, Day 120-180, and Day 330-420 unaided at a distance of 5 meters (m) using a chart. VA was measured in decimal, with 1.0 decimal corresponding to 20/20 Snellen. A higher numeric value represents better visual acuity.
Time Frame: Baseline (preoperative), Day 1-2, Day 7-14, Day 30-60, Day 120-180, Day 330-420
Population: This analysis population includes all implanted subjects.
Measure: Number; unit: participants
Groups:
- Preoperative; Day 1-2; Day 7-14; Day 30-60; Day 120-180; Day 330-420: AcrySof® IQ ReSTOR® +2.5 D Multifocal IOL Model SN6AD2
Arm/Group | Preoperative | Day 1-2 | Day 7-14 | Day 30-60 | Day 120-180 | Day 330-420
Number analyzed (Participants) | 64 | 64 | 64 | 64 | 64 | 63
participants
  First Eye worse than 0.5 decimal | 48 | 3 | 1 | 0 | 0 | 0
  First Eye 0.5 to less than 0.7 decimal | 9 | 9 | 6 | 9 | 7 | 6
  First Eye 0.7 to less than1.0 decimal | 6 | 22 | 17 | 19 | 20 | 13
  First Eye 1.0 decimal or better | 1 | 30 | 40 | 36 | 37 | 44
  Second Eye worse than 0.5 decimal | 49 | 7 | 1 | 0 | 0 | 0
  Second Eye 0.5 to less than 0.7 decimal | 5 | 7 | 8 | 7 | 6 | 3
  Second Eye 0.7 to less than 1.0 decimal | 8 | 21 | 17 | 21 | 17 | 22
  Second Eye 1.0 decimal or better | 2 | 29 | 38 | 36 | 41 | 38
  Binocular worse than 0.5 decimal | NA — Not Assessed | NA — Not Assessed | NA — Not Assessed | 0 | 0 | 0
  Binocular 0.5 to less than 0.7 decimal | NA — Not Assessed | NA — Not Assessed | NA — Not Assessed | 2 | 0 | 1
  Binocular 0.7 to less than 1.0 decimal | NA — Not Assessed | NA — Not Assessed | NA — Not Assessed | 14 | 14 | 7
  Binocular 1.0 decimal or better | NA — Not Assessed | NA — Not Assessed | NA — Not Assessed | 48 | 50 | 55

2. Primary Outcome: Uncorrected Decimal VA (50 cm)
Description: VA was tested monocularly at all visits and binocularly at Day 30-60, Day 120-180, and Day 330-420 unaided at a distance of 50 centimeters (cm) using a chart. VA was measured in decimal, with 1.0 decimal corresponding to 20/20 Snellen. A higher numeric value represents better visual acuity.
Time Frame: Baseline (preoperative), Day 1-2, Day 7-14, Day 30-60, Day 120-180, Day 330-420
Population: This analysis population includes all implanted subjects.
Measure: Number; unit: participants
Arm/Group | Preoperative | Day 1-2 | Day 7-14 | Day 30-60 | Day 120-180 | Day 330-420
Number analyzed (Participants) | 64 | 64 | 64 | 64 | 64 | 63
participants
  First Eye worse than 0.4 decimal | 49 | 12 | 6 | 4 | 5 | 2
  First Eye 0.4 decimal or better | 15 | 52 | 58 | 60 | 59 | 61
  Second Eye worse than 0.4 decimal | 44 | 11 | 4 | 3 | 5 | 3
  Second Eye 0.4 decimal or better | 20 | 53 | 60 | 61 | 59 | 60
  Binocular worse than 0.4 decimal | NA — Not Assessed | NA — Not Assessed | NA — Not Assessed | 2 | 2 | 0
  Binocular 0.4 decimal or better | NA — Not Assessed | NA — Not Assessed | NA — Not Assessed | 62 | 62 | 63

3. Primary Outcome: Best Corrected Decimal VA (5 m)
Description: VA was tested monocularly at all visits and binocularly at Day 30-60, Day 120-180, and Day 330-420 with the participant's best spectacle correction at a distance of 5 m using a chart. VA was measured in decimal, with 1.0 decimal corresponding to 20/20 Snellen. A higher numeric value represents better visual acuity.
Time Frame: Baseline (preoperative), Day 1-2, Day 7-14, Day 30-60, Day 120-180, Day 330-420
Population: This analysis population includes all implanted subjects.
Measure: Number; unit: participants
Arm/Group | Preoperative | Day 1-2 | Day 7-14 | Day 30-60 | Day 120-180 | Day 330-420
Number analyzed (Participants) | 64 | 64 | 64 | 64 | 64 | 63
participants
  First Eye worse than 0.5 decimal | 22 | 0 | 0 | 0 | 0 | 0
  First Eye 0.5 to less than 0.7 decimal | 18 | 3 | 0 | 0 | 1 | 0
  First Eye 0.7 to less than 1.0 decimal | 10 | 14 | 3 | 3 | 2 | 4
  First Eye 1.0 decimal or better | 14 | 47 | 61 | 61 | 61 | 59
  Second Eye worse than 0.5 decimal | 15 | 0 | 0 | 0 | 0 | 0
  Second Eye 0.5 to less than 0.7 decimal | 11 | 0 | 0 | 0 | 0 | 0
  Second Eye 0.7 to less than 1.0 decimal | 17 | 17 | 3 | 2 | 1 | 2
  Second Eye 1.0 decimal or better | 21 | 47 | 61 | 62 | 63 | 61
  Binocular worse than 0.5 decimal | NA — Not Assessed | NA — Not Assessed | NA — Not Assessed | 0 | 0 | 0
  Binocular 0.5 to less than 0.7 decimal | NA — Not Assessed | NA — Not Assessed | NA — Not Assessed | 0 | 0 | 0
  Binocular 0.7 to less than 1.0 decimal | NA — Not Assessed | NA — Not Assessed | NA — Not Assessed | 0 | 1 | 1
  Binocular 1.0 decimal or better | NA — Not Assessed | NA — Not Assessed | NA — Not Assessed | 64 | 63 | 62

4. Primary Outcome: Best Corrected Decimal VA (50 cm)
Description: VA was tested monocularly at all visits and binocularly at Day 30-60, Day 120-180, and Day 330-420 with the participant's best spectacle correction at a distance of 50 cm using a chart. VA was measured in decimal, with 1.0 decimal corresponding to 20/20 Snellen. A higher numeric value represents better visual acuity.
Time Frame: Baseline (preoperative), Day 1-2, Day 7-14, Day 30-60, Day 120-180, Day 330-420
Population: This analysis population includes all implanted subjects.
Measure: Number; unit: participants
Arm/Group | Preoperative | Day 1-2 | Day 7-14 | Day 30-60 | Day 120-180 | Day 330-420
Number analyzed (Participants) | 64 | 64 | 64 | 64 | 64 | 63
participants
  First Eye worse than 0.5 decimal | 22 | 7 | 1 | 0 | 0 | 1
  First Eye 0.5 to less than 0.7 decimal | 19 | 22 | 9 | 7 | 8 | 5
  First Eye 0.7 to less than 1.0 decimal | 12 | 30 | 38 | 39 | 35 | 32
  First Eye 1.0 decimal or better | 11 | 5 | 16 | 18 | 21 | 25
  Second Eye worse than 0.5 decimal | 11 | 4 | 0 | 0 | 1 | 1
  Second Eye 0.5 to less than 0.7 decimal | 19 | 22 | 6 | 3 | 4 | 4
  Second Eye 0.7 to less than 1.0 decimal | 17 | 28 | 43 | 42 | 37 | 28
  Second Eye 1.0 decimal or better | 17 | 10 | 15 | 19 | 22 | 30
  Binocular worse than 0.5 decimal | NA — Not Assessed | NA — Not Assessed | NA — Not Assessed | 0 | 0 | 0
  Binocular 0.5 to less than 0.7 decimal | NA — Not Assessed | NA — Not Assessed | NA — Not Assessed | 0 | 2 | 2
  Binocular 0.7 to less than 1.0 decimal | NA — Not Assessed | NA — Not Assessed | NA — Not Assessed | 29 | 26 | 17
  Binocular 1.0 decimal or better | NA — Not Assessed | NA — Not Assessed | NA — Not Assessed | 35 | 36 | 44

5. Primary Outcome: Distance-Corrected Decimal VA (50 cm)
Description: VA was tested monocularly at the preoperative, Day 30-60, Day 120-180, and Day 330-420 visits and binocularly at Day 30-60, Day 120-180, and Day 330-420 using a chart. Distance-corrected VA at 50 cm is the VA at 50 cm measured under a corrected condition in which best-corrected VA at 5 m was obtained. VA was measured in decimal, with 1.0 decimal corresponding to 20/20 Snellen. A higher numeric value represents better visual acuity.
Time Frame: Baseline (preoperative), Day 30-60, Day 120-180, Day 330-420
Population: This analysis population includes all implanted subjects.
Measure: Number; unit: participants
Arm/Group | Preoperative | Day 30-60 | Day 120-180 | Day 330-420
Number analyzed (Participants) | 64 | 64 | 64 | 63
participants
  First Eye worse than 0.4 decimal | 48 | 4 | 4 | 2
  First Eye 0.4 decimal or better | 16 | 60 | 60 | 61
  Second Eye worse than 0.4 decimal | 43 | 4 | 4 | 2
  Second Eye 0.4 decimal or better | 21 | 60 | 60 | 61
  Binocular worse than 0.4 decimal | NA — Not Assessed | 0 | 2 | 1
  Binocular 0.4 decimal or better | NA — Not Assessed | 64 | 62 | 62

6. Secondary Outcome: Uncorrected Decimal VA (1 m)
Description: VA was tested binocularly unaided at a distance of 1 m using a chart. VA was measured in decimal, with 1.0 decimal corresponding to 20/20 Snellen. A higher numeric value represents better visual acuity.
Time Frame: Day 120-180, Day 330-420
Population: This analysis population includes all implanted subjects.
Measure: Number; unit: participants
Arm/Group | Day 120-180 | Day 330-420
Number analyzed (Participants) | 64 | 63
participants
  Worse than 0.5 decimal | 0 | 0
  0.5 to less than 0.7 decimal | 8 | 3
  0.7 to less than 1.0 decimal | 20 | 22
  1.0 decimal or better | 36 | 38

7. Secondary Outcome: Distance Corrected Decimal VA (1 m)
Description: VA was tested binocularly using a chart. Distance-corrected VA at 1 m is the VA at 1 m measured under a corrected condition in which best-corrected VA at 5 m was obtained. VA was measured in decimal, with 1.0 decimal corresponding to 20/20 Snellen. A higher numeric value represents better visual acuity.
Time Frame: Day 120-180, Day 330-420
Population: This analysis population includes all implanted subjects.
Measure: Number; unit: participants
Arm/Group | Day 120-180 | Day 330-420
Number analyzed (Participants) | 64 | 63
participants
  Worse than 0.5 decimal | 3 | 0
  0.5 to less than 0.7 decimal | 4 | 3
  0.7 to less than 1.0 decimal | 24 | 26
  1.0 decimal or better | 33 | 34

8. Secondary Outcome: Uncorrected Decimal VA (40 cm)
Description: VA was tested binocularly unaided at a distance of 40 cm using a chart. VA was measured in decimal, with 1.0 decimal corresponding to 20/20 Snellen. A higher numeric value represents better visual acuity.
Time Frame: Day 120-180, Day 330-420
Population: This analysis population includes all implanted subjects.
Measure: Number; unit: participants
Arm/Group | Day 120-180 | Day 330-420
Number analyzed (Participants) | 64 | 63
participants
  Worse than 0.4 decimal | 3 | 2
  0.4 decimal or better | 61 | 61

9. Secondary Outcome: Distance Corrected Decimal VA (40 cm)
Description: VA was tested binocularly using a chart. Distance-corrected VA at 40 cm is the VA at 40 cm measured under a corrected condition in which best-corrected VA at 5 m was obtained. VA was measured in decimal, with 1.0 decimal corresponding to 20/20 Snellen. A higher numeric value represents better visual acuity.
Time Frame: Day 120-180, Day 330-420
Population: This analysis population includes all implanted subjects.
Measure: Number; unit: participants
Arm/Group | Day 120-180 | Day 330-420
Number analyzed (Participants) | 64 | 63
participants
  Worse than 0.4 decimal | 2 | 2
  0.4 decimal or better | 62 | 61

10. Secondary Outcome: Uncorrected Decimal VA at Best Distance
Description: VA was tested monocularly at all visits and binocularly at Day 30-60, Day 120-180, and Day 330-420 using a chart at the distance of best near vision (cm) as decided by the participant. VA was measured in decimal, with 1.0 decimal corresponding to 20/20 Snellen. A higher numeric value represents better visual acuity.
Time Frame: Baseline (preoperative), Day 1-2, Day 7-14, Day 30-60, Day 120-180, Day 330-420
Population: This analysis population includes all implanted subjects.
Measure: Number; unit: participants
Arm/Group | Preoperative | Day 1-2 | Day 7-14 | Day 30-60 | Day 120-180 | Day 330-420
Number analyzed (Participants) | 64 | 64 | 64 | 64 | 64 | 63
participants
  First Eye worse than 0.4 decimal | 52 | 13 | 6 | 4 | 5 | 3
  First Eye 0.4 decimal or better | 12 | 51 | 58 | 60 | 59 | 60
  Second Eye worse than 0.4 decimal | 48 | 14 | 6 | 4 | 3 | 5
  Second Eye 0.4 decimal or better | 16 | 50 | 58 | 60 | 61 | 58
  Binocular worse than 0.4 decimal | NA — Not Assessed | NA — Not Assessed | NA — Not Assessed | 2 | 2 | 1
  Binocular 0.4 decimal or better | NA — Not Assessed | NA — Not Assessed | NA — Not Assessed | 62 | 62 | 62

11. Secondary Outcome: Mean Best Distance (cm) for Uncorrected Decimal Near VA
Description: VA was tested monocularly at all visits and binocularly at Day 30-60, Day 120-180, and Day 330-420 unaided using a chart. The participant indicated the distance (cm) at which best near vision was attained.
Time Frame: Baseline (preoperative), Day 1-2, Day 7-14, Day 30-60, Day 120-180, Day 330-420
Population: This analysis population includes all implanted subjects. Here, "n" is the number of participants with non-missing values at the specific time point for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Preoperative | Day 1-2 | Day 7-14 | Day 30-60 | Day 120-180 | Day 330-420
Number analyzed (Participants) | 64 | 64 | 64 | 64 | 64 | 63
centimeters
  First Eye (n=45,64,64,64,64,63) | 40.5 (11.6) | 46.9 (5.2) | 47.3 (4.4) | 47.2 (3.8) | 47.3 (3.6) | 48.5 (3.6)
  Second Eye (n=47,64,64,64,64,63) | 39.8 (12.0) | 47.1 (3.8) | 46.9 (4.0) | 46.9 (3.7) | 47.5 (3.9) | 48.5 (3.7)
  Binocular (n=NA,NA,NA,64,64,63) | NA (NA) — Not Assessed | NA (NA) — Not Assessed | NA (NA) — Not Assessed | 47.0 (3.9) | 47.8 (3.6) | 48.9 (3.3)

12. Secondary Outcome: Mean Best Distance (cm) for Distance Corrected Decimal Near VA
Description: VA was tested monocularly at Day 1-2, Day 7-14, Day 30-60, Day 120-180, and Day 330-420 and binocularly at Day 30-60, Day 120-180, and Day 330-420 with the participant's best spectacle correction using a chart. The participant indicated the distance (cm) at which best near vision was attained.
Time Frame: Day 1-2, Day 7-14, Day 30-60, Day 120-180, Day 330-420
Population: This analysis population includes all implanted subjects.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Day 1-2 | Day 7-14 | Day 30-60 | Day 120-180 | Day 330-420
Number analyzed (Participants) | 64 | 64 | 64 | 64 | 63
centimeters
  First Eye | 48.2 (4.5) | 49.5 (4.4) | 48.6 (3.9) | 49.1 (3.3) | 49.4 (3.2)
  Second Eye | 48.2 (4.3) | 48.3 (3.5) | 48.5 (3.6) | 49.0 (3.3) | 49.2 (3.5)
  Binocular | NA (NA) — Not Assessed | NA (NA) — Not Assessed | 48.8 (3.9) | 48.8 (3.1) | 49.5 (3.1)

13. Secondary Outcome: Best Corrected Far (3 m) Contrast Sensitivity
Description: Far contrast sensitivity (ie, the ability to detect slight changes in luminance before they become indistinguishable) was assessed binocularly with the participant's best spectacle correction at a distance of 3 m using the Vector Vision CSV 1000 illuminated box (one site) and the Vision Contrast Test System (other site). Contrast sensitivity was assessed at spatial frequencies of 1.5, 3, 6, 12, and 18 cycles per degree (cpd). For CSV 1000, contrast sensitivity was not measured at spatial frequency 1.5 cpd because there was no option for this frequency. Raw scores were transformed to logMar (logarithm of the minimum angle of resolution) units. A higher numeric value represents better contrast sensitivity.
Time Frame: Day 120-180 from second eye implantation
Population: This analysis population includes all implanted subjects.
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- SN6AD2, as Measured With CSV-1000; SN6AD2, as Measured With VCTS: AcrySof® IQ ReSTOR® +2.5 D Multifocal IOL Model SN6AD2
Arm/Group | SN6AD2, as Measured With CSV-1000 | SN6AD2, as Measured With VCTS
Number analyzed (Participants) | 32 | 32
logMAR
  1.5 cpd | NA (NA) — Not an option for CSV-1000; therefore, not assessed. | 1.760 (0.227)
  3 cpd | 1.889 (0.130) | 2.047 (0.200)
  6 cpd | 2.026 (0.138) | 2.080 (0.187)
  12 cpd | 1.673 (0.186) | 1.800 (0.273)
  18 cpd | 1.176 (0.223) | 1.356 (0.244)

14. Secondary Outcome: Best Corrected Near (46 cm) Contrast Sensitivity
Description: Near contrast sensitivity (ie, the ability to detect slight changes in luminance before they become indistinguishable) was assessed binocularly with the participant's best spectacle correction at a distance of 46 cm using the Functional Acuity Contrast Test (FACT). Contrast sensitivity was assessed at spatial frequencies of 1.5, 3, 6, 12, and 18 cycles per degree (cpd). Raw scores were transformed to logMar units. A higher numeric value represents better contrast sensitivity.
Time Frame: Day 120-180 from second eye implantation
Population: This analysis population includes all implanted subjects.
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- SN6AD2: AcrySof® IQ ReSTOR® +2.5 D Multifocal IOL Model SN6AD2
Arm/Group | SN6AD2
Number analyzed (Participants) | 64
logMAR
  1.5 cpd | 1.825 (0.121)
  3 cpd | 1.933 (0.137)
  6 cpd | 1.739 (0.192)
  12 cpd | 1.311 (0.220)
  18 cpd | 0.856 (0.220)

15. Secondary Outcome: Mean Defocus Decimal VA (5 m)
Description: Defocus VA (an indicator of the expected range of vision with a presbyopia-correcting IOL) was tested binocularly with the participant's best spectacle correction at a distance of 5 m using a chart. Lenses of different spherical powers were placed in front of the eyes to produce varying levels of defocus. The VA at each spherical power was measured in decimal, with 1.0 decimal corresponding to 20/20 Snellen. A higher numeric value represents better visual acuity.
Time Frame: Day 120-180 from second eye implantation
Population: This analysis population includes all implanted subjects.
Measure: Mean (Full Range); unit: decimal
Arm/Group | SN6AD2
Number analyzed (Participants) | 64
decimal
  +2.00 | 0.44 [0.24 to 0.82]
  +1.50 | 0.65 [0.38 to 1.10]
  +1.00 | 0.85 [0.57 to 1.26]
  +0.50 | 1.11 [0.82 to 1.50]
  0.00 | 1.43 [1.16 to 1.76]
  -0.50 | 1.16 [0.90 to 1.49]
  -1.00 | 0.93 [0.68 to 1.28]
  -1.50 | 0.84 [0.62 to 1.15]
  -2.00 | 0.94 [0.67 to 1.31]
  -2.50 | 0.73 [0.51 to 1.05]
  -3.00 | 0.51 [0.32 to 0.80]
  -3.50 | 0.36 [0.22 to 0.58]
  -4.00 | 0.25 [0.15 to 0.41]
  -4.50 | 0.19 [0.11 to 0.30]
  -5.00 | 0.14 [0.08 to 0.24]

16. Secondary Outcome: Percentage of Participants With Positive Response, Stereoscopic Vision Test
Description: Stereopsis (the ability to perceive depth and 3-dimensional structure) was assessed binocularly under well-lit conditions at best distance using the Stereo Optical Company, Inc., Original Stereo Fly Test and polarized viewers. The participant was shown a series of symbols, with a positive response defined as correct identification of the 3-dimensional symbol. Responses were recorded for 3 symbols: Fly (easiest to perceive), animal, and circle (hardest to perceive).
Time Frame: Day 120-180 from second eye implantation
Population: This analysis population includes all implanted subjects.
Measure: Number; unit: percentage of participants
Arm/Group | SN6AD2
Number analyzed (Participants) | 64
percentage of participants
  House Fly | 100.0
  Animal | 93.8
  Circle | 85.9

17. Secondary Outcome: Percentage of Participants With Positive Response, Quality of Life Questions
Description: The participant completed a questionnaire, indicating (yes/no) if he/she experienced visual difficulty in every-day activities while not wearing spectacles. A positive response was defined as, "Yes=visual difficulty."
Time Frame: Day 120-180 from second eye implantation
Population: This analysis population includes all implanted subjects.
Measure: Number; unit: percentage of participants
Arm/Group | SN6AD2
Number analyzed (Participants) | 64
percentage of participants
  Reading small print, labels, telephone book | 89.1
  Reading a newspaper or a book | 81.3
  Reading dial plate of a wrist watch | 10.9
  Reading headline in a newspaper or book | 7.8
  Writing on papers or documents | 60.9
  Playing games such as chess, cards, mah-jongg | 1.6
  Drawing, sewing, knitting, or handiwork | 51.6
  Cooking | 15.6
  Watching TV | 3.1
  Seeing steps or stairs | 3.1
  Reading dial plate of clock or numbers on calendar | 3.1
  Recognizing people when they are close | 1.6
  Play table tennis, gate ball, tennis, golf, bowl | 4.7
  Reading a timetable in subway or train station | 6.3
  Reading plate of a bus or train coming | 1.6
  Reading traffic sign or shop sign | 1.6
  Seeing a PC screen | 42.2
  Seeing face in the mirror during makeup or shaving | 18.8
  Seeing distant blackboard or slide | 39.1

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of lens implantation for the duration of the study (May 9, 2012 to December 10, 2013). This reporting group includes all implanted subjects.
Description: An AE was defined as any untoward medical occurrence in a subject, user or other person regardless of whether or not the event had a causal relationship with the medical device or test procedures. Secondary surgical intervention (SSI) was also reported as an AE. AEs were collected as solicited comments and as observations by the study investigator.
Arm/Group | SN6AD2
Serious Adverse Events (participants affected / at risk) | 3/64
Other Adverse Events (participants affected / at risk) | 0/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SN6AD2 (N=64)
Uveitis (Eye disorders) | 1
Urinary Tract Infection (Infections and infestations) | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Intra-cerebral haemorrhage (Nervous system disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.